CLINICAL TRIAL: NCT01449084
Title: Immediate Pancreatic Duct Stent Removal Does Not Prevent Pancreatitis After Accidental Pancreatic Duct Cannulation - A Prospective Randomized Trial
Brief Title: Early Pancreatic Duct Stent Removal in Preventing Post-endoscopic Pancreatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nuovo Ospedale Civile S.Agostino Estense (Other)
Responsible Party: Principal Investigator, Rita Conigliaro, MD, Director, Head of Gastroenterology and Endoscopy Unit, NOCSAE, Nuovo Ospedale Civile S.Agostino Estense
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EPDSR
Record Dates: First submitted 2011-10-04; First posted 2011-10-07 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Acute Pancreatitis
Keywords: Pancreatic duct stenting; Post-endoscopic pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- early removal of pancreatic duct stent (Active Comparator): immediate removal of the pancreatic duct stent at the end of the ERCP procedure
  Interventions: Procedure: immediate stent removal
- leaving the stent in place (No Intervention): the pancreatic duct stent is left in place
  Interventions: Other: Leaving the stent in place

INTERVENTIONS:
Procedure: immediate stent removal — The stent used was a 5-Fr polyethylene duodenal pigtail pancreatic stent without an inner flange. The stent length was 4 or 5 cm (Zimmon stent, Cook Endoscopy, Winston-Salem, NC, USA): selection was based on the degree of flexion and the length of the Wirsung duct in the head of the pancreas.
  THE STENT WAS REMOVED AT THE END OF THE ERCP PROCEDURE
  Arms: early removal of pancreatic duct stent
Other: Leaving the stent in place — The stent used was a 5-Fr polyethylene duodenal pigtail pancreatic stent without an inner flange. The stent length was 4 or 5 cm (Zimmon stent, Cook Endoscopy, Winston-Salem, NC, USA): selection was based on the degree of flexion and the length of the Wirsung duct in the head of the pancreas.
  THE STENT WAS LEFT IN PLACE AT THE END OF THE ERCP PROCEDURE
  Arms: leaving the stent in place

SUMMARY:
Temporary pancreatic duct stent placement during endoscopic retrograde cholangiopancreatography (ERCP) has been recommended for post-endoscopic pancreatitis (PEP) prophylaxis in high risk patients, including those in whom accidental pancreatic duct cannulation has occurred. However, the optimal duration of stent placement remains an open question. The investigators aim is to assess if immediate stent removal is effective in the prevention of PEP after accidental pancreatic duct cannulation.

DETAILED DESCRIPTION:
Recent meta-analyses of randomized controlled trials confirmed that pancreatic stent placement after ERCP reduces the risk of PEP but the optimal duration of stent placement remains an open question. It has been suggested that in truly high-risk patients the pancreatic stent must be left in place for a minimum of 24 hours or more whereas in patients at lesser risk pancreatic duct drainage probably only needs to be maintained for a few hours or less. Leaving the stent in place at the end of the ERCP procedure carries the disadvantage of radiological follow-up until spontaneous dislodgment occurs or endoscopic removal is deemed timely; moreover, proximal migration has been reported, requiring endoscopic or even surgical removal. There is a paucity of data comparing immediate removal with spontaneous dislodgment in high-risk patients. In one study, significantly higher rates of PEP were detected in patients in whom a pancreatic stent was removed immediately at the end of the ERCP procedure than in those in whom the stent was left in place: unfortunately, only patients undergoing a precut sphincterotomy were evaluated in that study which was published only in abstract form. Therefore, it is still uncertain whether leaving a stent in place is more effective than immediate removal in preventing PEP in high-risk patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients in whom accidental pancreatic duct cannulation had occurred
* during guide wire directed ERCP

Exclusion Criteria:

* Patients who had undergone previous endoscopic papillectomy or sphincterotomy
* and those with an indwelled nasobiliary or nasopancreatic tube

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events, i.e. post-endoscopic pancreatitis | 24 h
  Post-endoscopic pancreatitis is defined as pancreatic pain and hyperamylasemia within 24 hours of the procedure and is assessed by a physician blinded to group assignment and to radiological surveillance findings. Pancreatic pain is defined as severe and persistent pain in the epigastric or periumbilical region. Hyperamylasemia is defined as an increase in the serum amylase level to greater than 3 times the upper normal limit. The pancreatitis is defined as mild, moderate, or severe according to the criteria proposed by Cotton et al. (GE 1991).

SECONDARY OUTCOMES:
Number of participants with proximal migration of the stent among those patients randomly assigned to leaving the stent in place. | 96 hours
  Radiological surveillance at 24-h intervals in order to detect proximal migration of the stent in the main pancreatic duct.

CONTACTS AND LOCATIONS:
Overall Officials: Rita Conigliaro, MD, Principal Investigator — Gastroenterologia - NOCSAE - Modena
Locations (1):
- Nuovo Ospedale Civile S. Agostino-Estense, Modena, Italy